CLINICAL TRIAL: NCT00457639
Title: Phase II Study of Cholic Acid for Hepatic Steatosis in Lipodystrophy Patients
Brief Title: Cholic Acid for Hepatic Steatosis in Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Abhimanyu Garg, PI, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 122010-032; FD003085
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hepatic Steatosis
Keywords: lipodystrophy
MeSH Terms: conditions — Fatty Liver; Lipodystrophy | interventions — Cholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholic Acid active capsules (Experimental): Cholic Acid weight based dose for 6 months double-blind
  Interventions: Drug: Cholic Acid
- Placebo for Cholic Acid (Placebo Comparator): Placebo for Cholic Acid for 6 months double-blind
  Interventions: Drug: Cholic Acid

INTERVENTIONS:
Drug: Cholic Acid — Capsules of active Cholic Acid or matching placebo, total dose is 15 mg/kg per day, maximum dose of 1500 mg per day, taken PO, BID.

SUMMARY:
To evaluate the efficacy and safety of cholic acid therapy in treating lipodystrophy patients with hepatic steatosis. This is a randomized, double-blind, placebo-controlled cross-over study.

DETAILED DESCRIPTION:
Lipodystrophies are rare disorders characterized by selective loss of adipose tissue and predisposition to develop insulin resistance and its associated metabolic complications such as dyslipidemia, diabetes mellitus and hepatic steatosis. Nonalcoholic hepatic steatosis or steatohepatitis caused by excessive accumulation of triglycerides in hepatocytes, in fact, is a common feature of these disorders. Often a cause for significant morbidity and even mortality in lipodystrophic patients, hepatic steatosis poses a significant therapeutic challenge. Recent insight into the role of primary bile acids, cholic acid and chenodeoxycholic acid, which are endogenous ligands for the farnesoid X receptor (FXR), in regulating hepatic triglyceride homeostasis offers new treatment options for hepatic steatosis. Cholic acid was shown to inhibit hepatic triglyceride accumulation by more than 50% in a mouse model of hepatic steatosis and hypertriglyceridemia. Cholic acid has been previously used to treat inborn errors of bile acid synthesis in children without any side effects. In other studies in adults, cholic acid has been reported to be well tolerated. Therefore, we propose to investigate a potentially safe therapeutic option for its efficacy in reducing hepatic steatosis in patients with lipodystrophies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lipodystrophies as diagnosed by clinical criteria.
* Hepatic steatosis (>5.6% hepatic triglyceride content) as demonstrated by 1H magnetic resonance spectroscopy.
* Age 6-70 years.
* Alcohol intake of less than 40 g per week.

Exclusion Criteria:

* Laboratory or other histologic findings highly suggestive of liver disease due to causes other than non-alcoholic steatohepatitis, such as chronic viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, biliary obstruction or genetic liver diseases such as Wilson's disease, hemochromatosis or alpha-1-antitrypsin deficiency.
* Treatment with drugs associated with steatohepatitis, e.g., corticosteroids, high dose estrogens, methotrexate, amiodarone, , sulfasalazine, or oxacillin in the 6 months prior to the study.
* Decompensated liver disease as evidenced by clinical features of hepatic failure (variceal bleeding, ascites, hepatic encephalopathy etc.) and laboratory investigations (prolonged prothrombin time, hypoalbuminemia, presence of esophageal varices etc.)
* Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study suggestive of liver cancer.
* Use of drugs which can potentially decrease hepatic steatosis during previous 3 months; ursodeoxycholic acid, high-dose vitamin E, betaine, acetylcysteine and choline. Thiazolidinediones are allowed if dose has been stable for 3 months prior to screening.
* Significant systemic or major illnesses other than liver disease, such as congestive heart failure, cerebrovascular disease, respiratory failure, renal failure (serum creatinine >2 mg/dL), acute pancreatitis, organ transplantation, serious psychiatric disease, and malignancy, that could interfere with the trial and adequate follow up.
* Acute medical illnesses precluding participation in the studies.
* Known HIV-infected patient.
* Current substance abuse.
* Pregnant or lactating women.
* Hematocrit of less than 30%. - History of weight loss during past 3 months.
* Patients on bile acid binding resins, cholestyramine, colestipol, colesevelam.
* Hypersensitivity or intolerance to CA or any components of its formulation

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Ahmad Z, Subramanyam L, Szczepaniak L, Simha V, Adams-Huet B, Garg A. Cholic acid for hepatic steatosis in patients with lipodystrophy: a randomized, controlled trial. Eur J Endocrinol. 2013 Apr 15;168(5):771-8. doi: 10.1530/EJE-12-0969. Print 2013 May. PMID 23447519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment December 2006 through April 2010. A total of 37 subjects were screened for this trial.
Groups:
- Cholic Acid Then Placebo: Cholic Acid for 6 months and then Placebo for six months in a double-blind, randomized fashion
- Placebo Then Cholic Acid: Placebo for 6 months and then Cholic Acid for 6 months in a double-blind, randomized fashion
Period: Intervention 1 (6 Months)
Arm/Group | Cholic Acid Then Placebo | Placebo Then Cholic Acid
Started | 9 (6 months on Cholic Acid and crossover to Placebo for 6 months) | 9 (6 months on Placebo and crossover to cholic acid for 6 months)
Completed | 6 (Number of Patients completing Cholic Acid Phase) | 7 (Number of patients completing Placebo Phase)
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — unrelated illness | 0 | 2
Period: Intervention 2 (6 Months)
Arm/Group | Cholic Acid Then Placebo | Placebo Then Cholic Acid
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Unrelated illness ineligible for MRS | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data is for all the patients enrolled
Groups:
- Characteristics of All Patients Enrolled: Participants who were randomized to receive either Cholic acid or Placebo
Arm/Group | Characteristics of All Patients Enrolled
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Hepatic TG (%) [Median (Full Range); unit: Fat/Fat+Water (%)] | 23.89 [6.1 to 60.3]
Serum Triglyceride [Median (Full Range); unit: mg/dL] | 389 [155 to 3455]

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Triglyceride (%)
Description: Measured by proton magnetic resonance spectroscopy (MRS)
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Fat/Fat+Water (%)
Groups:
- Cholic Acid: Cholic Acid 6 months .
- Placebo: Placebo for 6 months.
Arm/Group | Cholic Acid | Placebo
Number analyzed (Participants) | 13 | 15
Fat/Fat+Water (%) | 15.9 [10.5 to 26.5] | 14.8 [9.4 to 19]
Statistical Analysis 1: Comparison: Cholic Acid vs Placebo; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = 13.8, 95% CI 2-sided [-19.7 to 61.1]

2. Secondary Outcome: Serum Triglycerides
Time Frame: Months 6
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cholic Acid | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | 390 [233 to 595] | 340 [233 to 433]
Statistical Analysis 1: Comparison: Cholic Acid vs Placebo; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Final Values) = 11.4, 95% CI 2-sided [-17.7 to 50.8]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Diarrhea: Increased frequency of passing stool
Groups:
- Cholic Acid: Cholic Acid for 6 months
Arm/Group | Cholic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 5/14 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholic Acid (N=14) | Placebo (N=15)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — One patient developed gastroenteritis requiring intravenous fluids
Flu Like Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Flu like symptoms with vomiting and diarrhea.
Heart Failure (Cardiac disorders) | 0 (0) | 1 (4) — Fluid accumulation due to hear failure
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0) — Two patients developed diarrhea and excessive flatus while taking Cholic Acid. Their symptoms resolved after reducing the dosage. Three other patients reported mild diarrhea which subsided within one to two weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes